CLINICAL TRIAL: NCT05821972
Title: Nebulized Dexmedetomidine Combined With Ketamine Versus Nebulized Dexmedetomidine to Induce Preoperative Sedation and Attenuate Emergence Agitation in Children Undergoing Cleft Palate Repair Surgeries
Brief Title: Nebulized Dexmedetomidine Combined With Ketamine Versus Nebulized Dexmedetomidine for Cleft Palate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, FATMA NABIL AHMED MOHAMED, Clinical Supervisor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dexmedetomidine Ketamine
Record Dates: First submitted 2023-04-03; First posted 2023-04-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sedation; Emergence Delirium
Keywords: dexmedetomidine; Ketamine; Nebulization; Cleft palate; Sedation; Emergence delirium
MeSH Terms: conditions — Emergence Delirium; Cleft Palate | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized dexmedetomidine and ketamine (Experimental): Pre-operative nebulization of dexmedetomidine and ketamine
  Interventions: Drug: Nebulization of dexmedetomidine and ketamine
- Nebulized dexmedetomidine (Active Comparator): Pre-operative nebulization of dexmedetomidine
  Interventions: Drug: Nebulization of dexmedetomidine

INTERVENTIONS:
Drug: Nebulization of dexmedetomidine and ketamine — Pre-operative nebulization of dexmedetomidine and ketamine
  Arms: Nebulized dexmedetomidine and ketamine
Drug: Nebulization of dexmedetomidine — Pre-operative nebulization of dexmedetomidine
  Arms: Nebulized dexmedetomidine

SUMMARY:
To compare the efficacy of the pre-operative nebulization of a combination of dexmedetomidine and ketamine versus nebulization of dexmedetomidine alone for sedation and prevention of emergence delirium in children undergoing cleft palate repair surgeries.

DETAILED DESCRIPTION:
Cleft palate is a common congenital anomaly. The American cleft palate-craniofacial Association recommends that primary cleft palate repair should be ideally performed between 12-18 months after birth.

The pre-operative period is quite distressing for children due to parental separation, application of face mask for induction of anaesthesia, fear of needles and unfamiliar faces. Pre-operative Anxiety is associated with adverse outcomes via elevation of stress markers, promoting fluctuations in hemodynamic, and negatively impacting postoperative recovery. There is a growing interest in the use of dexmedetomidine, a highly selective alpha-2 adrenergic agonist, for paediatric premedication. Ketamine may attenuate dexmedetomidine-induced bradycardia and hypotension and accelerate the onset of sedation with no respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) physical status I & II who will be scheduled for cleft palate repair surgeries

Exclusion Criteria:

* Parent refusal
* Allergy to the study drugs
* Suspected difficult airway
* Patients with endocrine, renal, hepatic, and cardiac pathology
* Psychiatric diseases
* Asthmatic patients.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
University of Michigan Sedation Scale (UMSS) | Pre-operative
  It ranges from 0 = awake, alert to 4 = unarousable

SECONDARY OUTCOMES:
Parental Separation using the Parenteral Separation Anxiety Scale (PSAS) | Pre-operative
  It ranges from 1 = easy separation to 4 = crying and clinging to parents. Higher score means a worse outcome.
Watcha scale for emergence delirium | Postoperatively, up to 2 hours starting from arrival to the post-anesthesia care unit.
  It ranges from 1= calm to 4 = agitated

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt